CLINICAL TRIAL: NCT00279955
Title: Program to Access and Review Trending Information and Evaluate Correlation to Symptoms in Patients With Heart Failure
Brief Title: PARTNERS HF: Program to Access and Review Trending Information and Evaluate Correlation to Symptoms in Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 235
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure, Congestive; Implantable Cardioverter-Defibrillators
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy Device — Patients with an ICD indication, a CRT indication and symptomatic heart failure who are implanted with a Cardiac Resynchronization Therapy Device.

SUMMARY:
The purpose of this study is to determine the value of diagnostic data obtained from Medtronic implantable cardioverter defibrillators (ICDs) with cardiac resynchronization therapy (CRT) to evaluate cardiovascular and heart failure related adverse events and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the ICD indications
* Patients with Class III or IV heart failure.
* Patients receiving or who received a Medtronic CRT ICD within the previous 3 months.
* Patient must sign and date informed consent, and be 18 years of age or greater.
* Patient must be available for follow up visits, and be willing and able to comply with study protocol.

Exclusion Criteria:

* Patient with acute myocardial infarction (MI), coronary artery bypass graft surgery (CABG) or percutaneous coronary angioplasty (PTCA)/stent within the last month.
* Patient with a mechanical right heart valve.
* Patient with chronic (permanent) atrial arrhythmias.
* Patient with life expectancy of less than 12 months.
* Patient with status post heart transplant
* Patient undergoing kidney dialysis
* Patients enrolled in a concurrent study that may confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a specified Medtronic Implantable Cardiac Resynchronization Therapy Defibrillator device where informed consent and/or authorization to use and disclose health information permission has been granted.
Sampling Method: Non-Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Whellan, MD, Principal Investigator — Jefferson Heart Institute
Locations (93):
- United States (93):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Loma Linda, California
  - San Diego, California
  - Denver, Colorado
  - Guilford, Connecticut
  - Bradenton, Florida
  - Fort Lauderdale, Florida
  - Key Largo, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Orlando, Florida
  - Palm Beach Gardens, Florida
  - Pensacola, Florida
  - Safety Harbor, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Evanston, Illinois
  - Maywood, Illinois
  - Merrionette Park, Illinois
  - Rockford, Illinois
  - Springfield, Illinois
  - Winfield, Illinois
  - Topeka, Kansas
  - Wichita, Kansas
  - Edgewood, Kentucky
  - Florence, Kentucky
  - Louisville, Kentucky
  - Covington, Louisiana
  - Monroe, Louisiana
  - Portland, Maine
  - Salisbury, Maryland
  - Takoma Park, Maryland
  - Grand Rapids, Michigan
  - Marquette, Michigan
  - Petoskey, Michigan
  - Traverse City, Michigan
  - Minneapolis, Minnesota
  - Saint Cloud, Minnesota
  - St Louis, Missouri
  - Missoula, Montana
  - Las Vegas, Nevada
  - Manchester, New Hampshire
  - Cherryhill, New Jersey
  - Ridgewood, New Jersey
  - Sewell, New Jersey
  - New York, New York
  - The Bronx, New York
  - West Islip, New York
  - Williamsville, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Elyria, Ohio
  - Lakewood, Ohio
  - Mayfield Heights, Ohio
  - Westlake, Ohio
  - Medford, Oregon
  - Camp Hill, Pennsylvania
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wormleysburg, Pennsylvania
  - York, Pennsylvania
  - Pawtucket, Rhode Island
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Spartanburg, South Carolina
  - Sioux Falls, South Dakota
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Fairfax, Texas
  - Fort Worth, Texas
  - Lubbock, Texas
  - Burlington, Vermont
  - Lynchburg, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Kirkland, Washington
  - Green Bay, Wisconsin
  - Madison, Wisconsin

REFERENCES:
- [Derived] Whellan DJ, Ousdigian KT, Al-Khatib SM, Pu W, Sarkar S, Porter CB, Pavri BB, O'Connor CM; PARTNERS Study Investigators. Combined heart failure device diagnostics identify patients at higher risk of subsequent heart failure hospitalizations: results from PARTNERS HF (Program to Access and Review Trending Information and Evaluate Correlation to Symptoms in Patients With Heart Failure) study. J Am Coll Cardiol. 2010 Apr 27;55(17):1803-10. doi: 10.1016/j.jacc.2009.11.089. PMID 20413029
- [Derived] Whellan DJ, O'Connor CM, Ousdigian KT, Lung TH; PARTNERS HF Study Investigators. Rationale, design, and baseline characteristics of a Program to Assess and Review Trending INformation and Evaluate CorRelation to Symptoms in Patients with Heart Failure (PARTNERS HF). Am Heart J. 2008 Nov;156(5):833-9, 839.e2. doi: 10.1016/j.ahj.2008.06.036. Epub 2008 Sep 23. PMID 19061695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1024 subjects were enrolled in the study from 21 JUN 2004 through 14 FEB 2007 from 100 centers in US. Follow-up data collection ended on 06 MAR 2008.
Pre-assignment Details: 23 of 1024 subjects exited prior to successful implant due to not meeting in/exclusion criteria, unsucessful implants, missing informed consent form etc. Of the remaining 1001 subjects, 643 subjects had been followed longer than 6 months and had the OptiVol feature save-to-disk data available. Those 643 subjects were used for analyzing objectives.
Groups:
- At Least 1 OptiVol Fluid Index > 100 During DREP: All subjects who were followed longer than 6 months and had OptiVol fluid index crossing 100 during DREP. An OptiVol index > 100 indicates potential fluid retention in the lungs. DREP: Diagnostic Risk Evaluation Period which is defined from consent date or implant date to 6 month visit.
- No OptiVol Fluid Index > 100 During DREP: All subjects who were followed longer than 6 months and never had OptiVol Fliud index crossing 100 during DREP. DREP: Diagnostic Risk Evaluation Period which is defined from consent date or implant date to 6 month visit.
- No OptiVol Measurement: All subjects either who were not followed for at least 6 months, or didn't have OptiVol Fluid Index measurements available.
Period: Overall Study
Arm/Group | At Least 1 OptiVol Fluid Index > 100 During DREP | No OptiVol Fluid Index > 100 During DREP | No OptiVol Measurement
Started | 157 | 486 | 358
Completed | 157 | 486 | 358 (They are still counted as completes, though they are never used for the analyses of objectives.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | At Least 1 OptiVol Fluid Index > 100 During DREP | No OptiVol Fluid Index > 100 During DREP | No OptiVol Measurement | Total
Number analyzed (Participants) | 157 | 486 | 358 | 1001
Age Continuous [Mean (Standard Deviation); unit: years] | 68.8 (11.0) | 68.2 (10.6) | 68.5 (11.0) | 68.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 163 | 109 | 317
  Male | 112 | 323 | 249 | 684
Region of Enrollment [Number; unit: participants]
  United States | 157 | 486 | 358 | 1001

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Heart Failure (HF) Related Adverse Event (AE)
Description: Number of participates with HF realted adverse event will be reported. Time to the first HF related Adverse event in the "Follow-up Period" from the 6-month visit to the 12-month visit is compared between two risk groups. The goal was to test if there is a significant difference in time to first HF-related adverse event between two groups. A heart failure related (HF-related) adverse event is defined as an adverse event that results in a subject's worsening HF or related to the heart's inability to meet the metabolic demands of the body.
Time Frame: From 6 month to the 12 month visit
Population: Of the 1001 subjects meeting inclusion and exclusion criteria, 643 subjects had been followed longer than 6 months and had the OptiVolTM feature save-to-disk data available. Those 643 subjects were included in this analysis.
Measure: Number; unit: participants
Arm/Group | At Least 1 OptiVol Fluid Index > 100 During DREP | No OptiVol Fluid Index > 100 During DREP
Number analyzed (Participants) | 157 | 486
participants | 29 | 50
Statistical Analysis 1: Comparison: At Least 1 OptiVol Fluid Index > 100 During DREP vs No OptiVol Fluid Index > 100 During DREP; Test type: Superiority or Other; p = 0.0119, Regression, Cox; Cox Proportional Hazard = 2.07, 95% CI 2-sided [1.17 to 3.67], Standard Deviation 0.292 — The estimated parameter in a Cox regression model was adjusted by age, gender, New York Heart Association (NYHA) class at 6 month visit, Angiotensin Converting Enzyme (ACE)/Angiotensin Receptor Blocker (ARB) at 6 months, and Diuretics at 6 month

2. Secondary Outcome: Occurrence of Heart Failure (HF) Related Healthcare Utilization (HU)
Description: Number of participates with HF realted healthcare utilization will be reported. Time to the first HF-related healthcare utilization in the "Follow-up Period" from the 6-month visit to the 12-month visit is compared between two risk groups. The goal was to test if there is a significant difference in time to first HF-related healthcare utilization between two groups. A heart failure related (HF-related) healthcare utilization is defined as unscheduled office visits, hospitalizations, urgent care visits, and emergency room visits which is resulted by heart failure related adverse event.
Time Frame: 6 month to the 12 month visit
Measure: Number; unit: participants
Arm/Group | At Least 1 OptiVol Fluid Index > 100 During DREP | No OptiVol Fluid Index > 100 During DREP
Number analyzed (Participants) | 157 | 486
participants | 22 | 35
Statistical Analysis 1: Comparison: At Least 1 OptiVol Fluid Index > 100 During DREP vs No OptiVol Fluid Index > 100 During DREP; Test type: Superiority or Other; p = 0.0185, Regression, Cox; Cox Proportional Hazard = 1.90, 95% CI 2-sided [1.11 to 3.27], Standard Deviation 0.277 — The estimated parameter in a Cox regression model was adjusted by age, gender, NYHA class at 6 month visit, ACE/ARB at 6 months, and and at least one day where CRT pacing <90% in last 21 days of DREP

3. Secondary Outcome: Occurrence of Heart Failure (HF) Related Pulmonary Congestion Event (PCE)
Description: Number of participates with HF related pulmonary congestion event will be reported. Time to the first HF related pulmonary cogestion event in the "Follow-up Period" from the 6-month visit to the 12-month visit is compared between two risk groups to see if there is significant difference. A HF related pulmonary congestion event is defined as hospitalization with signs and/or symptoms of pulmonary congestion, or outpatient treatment with IV diuretics due to exacerbation of HF with signs and/or symptoms of pulmonary congestion.
Time Frame: 6 month to the 12 month visit
Measure: Number; unit: participants
Arm/Group | At Least 1 OptiVol Fluid Index > 100 During DREP | No OptiVol Fluid Index > 100 During DREP
Number analyzed (Participants) | 157 | 486
participants | 17 | 28
Statistical Analysis 1: Comparison: At Least 1 OptiVol Fluid Index > 100 During DREP vs No OptiVol Fluid Index > 100 During DREP; Test type: Superiority or Other; p = 0.0578, Regression, Cox; Hazard Ratio (HR) = 1.80, 95% CI 2-sided [0.98 to 3.31], Standard Deviation 0.311 — A Cox regression model has been used here, and the estimated parameter has been adjusted by including covariates age, gender, and NYHA class at 6 months

ADVERSE EVENTS:
Time Frame: Those adverse events were collected during the study (0 to 12 month follow-up).
Description: All adverse events which resulted in hospitalization are listed as serious adverse events.
Arm/Group | At Least 1 OptiVol Fluid Index > 100 During DREP | No OptiVol Fluid Index > 100 During DREP | No OptiVol Measurement
Serious Adverse Events (participants affected / at risk) | 84/157 | 114/486 | 99/358
Other Adverse Events (participants affected / at risk) | 75/157 | 172/486 | 96/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | At Least 1 OptiVol Fluid Index > 100 During DREP (N=157) | No OptiVol Fluid Index > 100 During DREP (N=486) | No OptiVol Measurement (N=358)
Atrial fibrillation (General disorders) | 2 (2) | 10 (11) | 4 (4)
Atrial flutter (General disorders) | 1 (1) | 5 (6) | 1 (1)
Atrial tachycardia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiomyopathy (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pressure/tightness (General disorders) | 0 (0) | 3 (3) | 3 (3)
Chronic obstructive pulmonary disease (General disorders) | 1 (1) | 3 (3) | 0 (0)
Dehydration (General disorders) | 0 (0) | 3 (3) | 1 (1)
Dizziness (General disorders) | 0 (0) | 2 (2) | 2 (2)
Dyspnea/Shortness of breath (General disorders) | 12 (17) | 21 (29) | 18 (21)
Fatigue, tiredness (General disorders) | 1 (1) | 1 (1) | 1 (1)
Heart failure decompensation (General disorders) | 24 (35) | 22 (24) | 24 (30)
Hypertension (General disorders) | 0 (0) | 1 (2) | 0 (0)
Hypotension (General disorders) | 3 (3) | 4 (4) | 1 (1)
Ischemic heart disease (General disorders) | 0 (0) | 1 (1) | 0 (0)
Near (pre) syncope (General disorders) | 1 (1) | 0 (0) | 1 (1)
PVC's (General disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysymal nocturnal dyspnea (General disorders) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (General disorders) | 1 (1) | 3 (3) | 0 (0)
Peripheral edema (General disorders) | 0 (0) | 0 (0) | 4 (4)
Peripheral vascular disease (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Pleural effusion (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (General disorders) | 2 (2) | 1 (1) | 2 (2)
Renal failure (General disorders) | 1 (1) | 0 (0) | 1 (1)
Shoulder pain/discomfort (General disorders) | 1 (2) | 0 (0) | 0 (0)
Syncope (General disorders) | 1 (1) | 4 (4) | 2 (2)
Thrombosis (General disorders) | 1 (1) | 2 (2) | 1 (1)
Vascular heart disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Ventricular tachycardia (General disorders) | 5 (6) | 8 (9) | 2 (2)
Wheezing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening cough (General disorders) | 1 (1) | 1 (1) | 0 (0)
xOther Intrinsic Rhythm/Conduction Codes (General disorders) | 1 (1) | 1 (1) | 1 (1)
yOther patient disease/condition codes (General disorders) | 0 (0) | 1 (1) | 2 (3)
zAll "Other" codes (General disorders) | 23 (27) | 13 (14) | 19 (19)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | At Least 1 OptiVol Fluid Index > 100 During DREP (N=157) | No OptiVol Fluid Index > 100 During DREP (N=486) | No OptiVol Measurement (N=358)
Arm/hand swelling (General disorders) | 0 (0) | 2 (2) | 1 (1)
Atrial fibrillation (General disorders) | 3 (5) | 6 (6) | 6 (6)
Atrial flutter (General disorders) | 0 (0) | 3 (3) | 2 (2)
Atrial tachycardia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pressure/tightness (General disorders) | 0 (0) | 3 (5) | 1 (1)
Chronic obstructive pulmonary disease (General disorders) | 2 (2) | 2 (3) | 1 (1)
Dehydration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (General disorders) | 4 (4) | 12 (12) | 4 (8)
Dyspnea/Shortness of breath (General disorders) | 23 (30) | 39 (43) | 19 (23)
Fatigue, tiredness (General disorders) | 3 (3) | 16 (16) | 3 (3)
Heart failure decompensation (General disorders) | 6 (7) | 8 (8) | 4 (6)
Hypertension (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (General disorders) | 3 (3) | 2 (2) | 4 (4)
Near (pre) syncope (General disorders) | 2 (2) | 2 (3) | 3 (3)
PVC's (General disorders) | 0 (0) | 2 (2) | 0 (0)
Palpitations (General disorders) | 1 (1) | 5 (5) | 1 (1)
Paroxysymal nocturnal dyspnea (General disorders) | 1 (3) | 4 (4) | 1 (1)
Pericardial effusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral edema (General disorders) | 6 (7) | 16 (20) | 10 (10)
Peripheral vascular disease (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (General disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 7 (7) | 2 (2)
Thrombosis (General disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular fibrillation (General disorders) | 0 (0) | 7 (7) | 5 (5)
Ventricular tachycardia (General disorders) | 2 (2) | 3 (8) | 6 (9)
Wheezing (General disorders) | 1 (1) | 2 (2) | 0 (0)
xOther Intrinsic Rhythm/Conduction Codes (General disorders) | 1 (1) | 1 (1) | 2 (2)
yOther Patient Disease/Conduction Codes (General disorders) | 1 (1) | 8 (8) | 4 (4)
zAll "Other" Codes (General disorders) | 12 (19) | 17 (20) | 12 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigation Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication. PI's may not publish single-site data until the main multi-site publication has occurred.